CLINICAL TRIAL: NCT04801732
Title: The Effect of Mulligan Thoracic Sustained Natural Apophyseal Glides on Sub-acromial Impingement Syndrome.
Brief Title: The Effect of Thoracic Mulligan Mobilization on Sub-acromial Impingement Syndrome
Acronym: SAIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Fatma Al-Zahraa Ahmad Alaa Aldin Mansour Abo-oof, physical therapist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Basic Science PT; faculty of physical therapy (Other: Cairo University)
Record Dates: First submitted 2021-03-07; First posted 2021-03-17 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Shoulder Impingement Syndrome
Keywords: SUBACROMIAL IMPINGEMENT SYNDROME; mulligan thoracic sustained natural apophyseal glides; Acromiohumeral distance or subacromial space
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized controlled study design were the recruited patients will randomly allocated into two groups control group and study group by Closed Envelope method of randomization. The treatment for all patients in both groups will conducted 3 times per week for one month .The study group (A): will receive SNAGS techniques on thoracic spine with traditional treatment consist of ice application, supervised exercises (stretching and strengthening exercise) and the study group(B) will receive only traditional treatment (ice or application and supervised exercise). All patients will be diagnosed as stage II according to Neer's classification recruited from orthopedic clinic from both sexes who met all the inclusion criteria and will be informed about the study procedure and signed the informed consent prepared for this study.
Who Masked: Participant
Masking Description: Patients will randomly assigned into two groups without being informed whether they are in the control or the study(experimental) group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mulligan group (Experimental): Patients in the study group will treated with SNAGS techniques on thoracic spine with traditional treatment consist of ice application, supervised exercises (stretching and strengthening exercise) for 3 times/week for one month.
  Interventions: Other: mulligan thoracic Sustained Natural Apophyseal Glides
- exercising group (Active Comparator): will receive only traditional treatment (ice application and supervised exercise ) for 3 times/week for one month.
  Interventions: Other: traditional treatments

INTERVENTIONS:
Other: mulligan thoracic Sustained Natural Apophyseal Glides — Extension Thoracic Sustained Natural Apophyseal Glides :
  Patient position: The patient sits astride the end of the table with hands placed behind the neck to protract the scapulae allowing access to the mid thoracic spine for the therapist's hand.
  Therapist position: Therapist stands on their most efficient side for a centrally applied Sustained Natural Apophyseal Glides.
  Therapist grasp: The therapist's mobilizing hand (ulnar border) will apply a cephalad glide in line with the facet joint plane of the involved spinal level and the other arm holds the thoracic wall above the level to be mobilized.
  Traction is applied prior to glide, which is achieved by therapist knee extension
  Repetitions: Three sets of ten repetitions will be done after a trial for the patient to be familial with the technique.
  and traditional treatment.
  Arms: mulligan group
Other: traditional treatments — includes: Ice pack and Pendulum exercise and shoulder range of motion (elevation, depression, flexion, abduction, rotations).Stretching exercise for internal rotators and posterior capsule.
  Strengthening exercise will be isometric in nature include external shoulder rotators, internal rotators, biceps, deltoid, and scapular stabilizers (rhomboids, trapezius, serratus anterior, Latissimus Dorsi , and pectoralis major muscles).
  Arms: exercising group

SUMMARY:
This study was conducted to investigate the effect of mulligan thoracic sustained natural apophyseal glide on patients diagnosed as sub acromial impingement syndrome and its effect on shoulder range of motion, pain, function and disability of affected shoulder joint and size of sub acromial space, Half of the patients will treated with traditional treatment and mulligan thoracic SNAGS technique, while the other half will treated with traditional treatment only.

DETAILED DESCRIPTION:
Forty patients with sub-acromial impingement syndrome will participate in this study. Intervention for the both group consisted of 12 session (3 times per week ) for one month. Subjects will be divided randomly and allocated into two groups , study group will received supervised exercise and mulligan thoracic SNAGS technique and the control group will received supervised exercise (stretching and strengthening exercises). both group will assessed by x ray to measure sub-acromial space , visual analogue scale for pain , The Shoulder Pain and Disability Index for shoulder function and goniometer for shoulder flexion, abduction ,external and internal rotation range of motion before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients referred as sub-acromial impingement syndrome (stage 2) according to neer's classification.
2. Have +ve Neer's sign, +ve Hawkins and Kennedy test and +ve Empty and full can tests.
3. selected from both genders.
4. Aged from 25 to 40 years old.
5. Have restricted thoracic extension motion ( +ve occiput to wall test).

Exclusion Criteria:

1. History of shoulder adhesive capsulitis
2. Rotator cuff tendon tear/rupture (stage 3).
3. Shoulder dislocation, subluxation and fractures.
4. History of cervical, shoulder, upper back surgery.
5. Any spinal deformities such as scoliosis, kyphosis and rounded shoulder.
6. Diabetes mellitus.
7. Radiculopathy.
8. History of breast cancer.
9. Previous stroke or Shoulder hand syndrome.
10. Ligamentous Laxity.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Pain by Visual analogue scale | changes from baseline to before treatment and changes before treatment to immediately after treatment
  the patient asked to choose from scale from zero (no pain) to 10 (worst pain) to detect his/her intensity of pain.
Range of motion of shoulder joint by universal goniometer. | changes from baseline to before treatment and changes before treatment to immediately after treatment
  for flexion stationary Arm of the goniometer was aligned with the lateral border of the scapula (mid axillary arm), and the moving arm was aligned with the humerus.
  for abduction the fulcrum was placed at the mid point of the posterior aspect of the glenohumeral joint, stationary arm was parallel to the trunk, and the moving arm was parallel to the longitudinal axis of the humerus. for internal and external rotation patient was in supine with the hips and knees flexed approximately 45°.The tested arm was supported on the table in 90° of abduction, elbow flexed 90°, and the wrist in neutral position.
  the fulcrum was placed on the olecranon, stationary arm Placed perpendicular to the floor, and the moving arm parallel with the forearm.
Shoulder pain and disability index | changes from baseline to before treatment and changes before treatment to immediately after treatment
  the patients will asked to answer the questions on index . And then creating a percentage of pain and disability with higher scores indicating more severe limitation. The means of the two subscales are averaged to produce a total score ranging from 0 (best) to 100 (worst).
  Minimum Detectable Change (90% confidence) = 13 points
The sub-acromial space by radiograph X ray | changes from baseline to before treatment and changes before treatment to immediately after treatment
  measure the size of sub-acromial space

CONTACTS AND LOCATIONS:
Overall Officials: Shimaa T Abu EL-Kasem, PhD, Principal Investigator — Cairo University
Locations (1):
- faculty of physical therapy - Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
These data are case sensitive and considered confidential regarding my supervisors' and study directors' opinion, So, upon their request i prefer to not share individual participant data with other researchers